# Information and consent "Preoperative measurement of abdominal circumference as a predictor of difficult spinal anesthesia and maternal hypotension during caesarian section"

# PATIENT INFORMATION AND CONSENT LETTER FOR PARTICIPATION IN MEDICAL RESEARCH

Research title: Validation of a study on abdominal perimeter measurement and caesarean section

Dear Madam,

We would like to invite you to participate in a clinical research study. This document explains what this study involves. Please take the time to read and understand this information, to think about your participation and to ask the doctor in charge of the study to explain anything you may not have understood.

#### I. PURPOSE OF THE STUDY:

To determine the threshold value of abdominal perimeter predictive of difficulty in performing spinal anesthesia for cesarean section and the occurrence of maternal arterial hypotension.

# II. EXPECTED BENEFITS

New, easy-to-assess clinical tool for optimizing spinal anesthesia technique with ultrasound and preventing maternal hypotension thus improving patient comfort and safety.

# III. STUDY PROCEDURE

Clinical data will be collected anonymously from your medical record, and the anesthesiologist will then measure your abdominal circumference, height, weight ,Body Mass Index, abdominal circumference in standing and sitting positions, and trunk length.

# IV. POTENTIAL RISKS

As this is a simple examination to be completed prior to your surgery, no adverse effects are expected and it will in no way affect the quality of your care. Answers are anonymous and no financial participation is expected.

#### V. CONFIDENTIALITY

All information concerning you collected during this work will be treated as confidential.

Only the people in charge of the study, and possibly the health authorities, will have access to this data. With the exception of these people - who will treat the information with the strictest respect for medical confidentiality - your anonymity will be preserved. The publication of the study results will not include any individual results, in compliance with the laws governing the processing of nominative data for health research purposes. If you have any questions during your participation in this study, please contact the doctors in charge of the study.

You are free to accept or refuse to participate in this study. This will not affect the quality of care you receive. Thank you for taking the time to read this newsletter. If you agree to participate in this research, we invite you to sign the enclosed consent form.

# **CONSENT FORM**

| I, the undersigned(Name and surname), agree to |
|---|
| participate in the study on abdominal perimeter measurement and caesarean section. |
| The objectives and modalities of the study have been clearly explained to me by the |
| investigators. |
| I have read and understood the information sheet provided to me. |
| I accept that the documents in my medical file relating to the study may be made available to |
| the persons in charge of the study and, if necessary, to the health authorities. With the |
| exception of these persons, who will handle the information in strict compliance with medical |
| secrecy, my anonymity will be preserved. |
| I understand that my participation in the study is voluntary. |
| I am free to accept or refuse to participate, and I am free to stop my participation at any time |
| during the study. This will not affect the quality of care I receive. |
| My consent does not relieve the organizers of this study of their responsibilities. I retain all |
| my rights guaranteed by law. |
| After discussing this matter and obtaining answers to all my questions, I freely and voluntarily |
| agree to take part in the research proposed to me. |
| Signed in Marrakech, |
| (Name and signature of patient) |
| Name and signature of investigator |

#### LETTRE D'INFORMATION ET DE CONSENTEMENT DESTINEE AUX PATIENTES

#### POUR PARTICIPATION A UNE RECHERCHE MEDICALE

Titre de la recherche : Validation d'une étude sur la mesure du périmètre abdominal et la césarienne

Madame,

Nous vous proposons de participer à une étude de recherche clinique. Cette lettre d'information vous détaille en quoi consiste cette étude. Vous pourrez prendre le temps pour lire et comprendre ces informations, de réfléchir à votre participation et pour demander au médecin responsable de l'étude de vous expliquer ce que vous n'aurez pas compris.

#### I. BUT DE L'ÉTUDE :

Déterminer la valeur seuil du périmètre abdominal prédictif de la difficulté de réalisation de la rachianesthésie pour césarienne et la survenue d'hypotension artérielle.

#### II. BÉNÉFICES ATTENDUS

Nouvel outil clinique facile d'évaluation permettant d'optimiser la technique de rachianesthésie avec l'échographie et la prévention de l'hypotension maternelle.

#### III. DÉROULEMENT DE L'ÉTUDE

Des données cliniques seront relevées à partir de votre dossier médical de façon anonyme, ensuite le médecin anesthésiste réanimateur prendra mesure de votre périmètre abdominal ne mesure de votre taille, poids (IMC) du périmètre abdominal en position debout et assise et de la longueur du tronc.

#### IV. RISQUES POTENTIELS

Aucun effet indésirable n'est attendu vu qu'il s'agit d'un simple questionnaire à remplir avant votre chirurgie, il n'affectera en rien la qualité de votre prise en charge. Les réponses sont anonymes et aucune participation financière n'est attendue.

# V. <u>CONFIDENTIALITE</u>

Toute information vous concernant recueillie pendant ce travail sera traitée de façon confidentielle.

Seuls les responsables de l'étude et éventuellement les autorités de Santé pourront avoir accès à ces données. A l'exception de ces personnes -qui traiteront les informations dans le plus strict respect du secret médical, votre anonymat sera préservé. La publication des résultats de l'étude ne comportera aucun résultat individuel conformément aux lois relatives au traitement des données nominatives ayant pour fin la recherche dans le domaine de la santé. Si vous avez des questions pendant votre participation à cette étude, vous pourrez contacter les médecins responsables de l'étude.

Vous êtes libre d'accepter ou de refuser de participer à cette étude. Cela n'influencera pas la qualité des soins qui vous seront prodigués. Nous vous remercions d'avoir pris le temps de lire cette lettre d'information. Si vous êtes d'accord pour participer à cette recherche, nous vous invitons à signer le formulaire de consentement cijoint.

# FORMULAIRE DE CONSENTEMENT

| Je soussignee |
|---|
| l'étude portant sur la mesure du périmètre abdominal et la césarienne. |
| Les objectifs et modalités de l'étude m'ont été clairement expliqués par les responsables de l'étude. |
| J'ai lu et compris la fiche d'information qui m'a été remise. |
| J'accepte que les documents de mon dossier médical qui se rapportent à l'étude puissent être accessibles aux |
| responsables de l'étude et éventuellement aux autorités de santé. A l'exception de ces personnes, qui traiteront |
| les informations dans le plus strict respect du secret médical, mon anonymat sera préservé. |
| J'ai bien compris que ma participation à l'étude est volontaire. |
| Je suis libre d'accepter ou de refuser de participer, et je suis libre d'arrêter à tout moment ma participation en cours d'étude. Cela n'influencera pas la qualité des soins qui me seront prodigués. |
| Mon consentement ne décharge pas les organisateurs de cette étude de leurs responsabilités. Je conserve tous mes droits garantis par la loi. |
| Après en avoir discuté et avoir obtenu la réponse à toutes mes questions, j'accepte librement et volontairement de participer à la recherche qui m'est proposée. |
| Fait à Marrakech, |
| le |
| Nom et signature de l'investigateur Signature du patient |

# نص المعلومات ونموذج موافقة المرضى للمشاركة في الأبحاث السريرية

# عنوان البحث

قياس محيط البطن قبل الجراحة كمؤشر لصعوبة التخدير الشوكي وانخفاض ضغط الدم لدى الأم أثناء الولادة" "القيصرية

سيداتي سادتي،

هذه النص يشرح تفاصيل هذه الدراسة نقترح عليك المشاركة في دراسة سريرية

# الهدف من الدراسة

يساعد في التقييم السابق للعمليات الجراحية والتحضير الأفضل لحدوث المضاعفات الفورية

# الفوائد المتوقعة

أداة سريرية لتقييم صعوبة التخدير النخاعي وحدوث انخفاض ضغط الدم الشرياني الأمومي

# تقديم الدراسة

سيتم جمع البيانات السريرية من ملفك الطبي دون الكشف عن هويتك ، ثم يجب عليك الإجابة على استبيان يتكون من 15 سؤالًا بمتوسط وقت استجابة يبلغ 3 دقائق. سيتم إرسال نفس الاستبيان إليك مرة أخرى في اليوم التالي للجراحة ، إما وجهاً لوجه أو عبر الهاتف ، حسب اختيارك.

# المخاطر المحتملة

لا يُتوقع حدوث آثار جانبية نظرًا لأن هذا استبيان بسيط يجب إكماله قبل الجراحة وبعدها ، فلن يؤثر بأي حال من الأحوال على جودة رعايتك. الموظفون المسؤولون عن الدراسة مستقلون عن فريق الرعاية الصحية الخاص بكولا يتوقع أي مشاركة مالية.

.

سرية المعلومات: سوف تعامل معلوماتك بسرية كاملة و لن يطلع على بياناتك سوى الباحث الرئيسي مع عدم ذكر الاسم و النسب .

حقوق المشارك: منحقكا لامتناع عنالمشاركة فيهذا البحثو فيهذها لحالة ستتلقب علاجكالمعتاد

# عندوجود استفسارلديك يمكنك الاتصال ب الباحث الرئيسى

شكرا لأخذ الوقت الكافي لقراءة هذه الرسالة الإخبارية. إذا وافقت على المشاركة في هذا البحث، فإننا ندعوك للتوقيع على نموذج الموافقة المرفق

# موافقة المريض

أنا الموقع أدناه ...... (الاسم واللقب) ،

يوافق على المشاركة في الدراسة المذكورة أعلاه

تم شرح أهداف وطرائق الدراسة بوضوح لي من قبل الدكتور

قرأت وفهمت ورقة المعلومات التي قدمت لي

أوافق على أن الوثائق الموجودة في ملفي الطبي المتعلقة بالدراسة قد تكون متاحة لقادة الدراسة وربما للسلطات الصحية. باستثناء هؤلاء الأشخاص ، الذين سيتعاملون مع المعلومات بأقصى درجات الاحترام للسرية الطبية ، سيتم الحفاظ على . هويتي

أفهم أن مشاركتي في الدراسة طوعية

أنا حر في قبول أو رفض المشاركة ، وأنا حر في أن أتوقف في أي وقت عن مشاركتي في الدراسة. هذا لن يؤثر على . جودة الرعاية التي سيتم تقديمها لي

موافقتي لا تعفى منظمي هذه الدراسة من مسؤولياتهم. أحتفظ بجميع حقوقي التي يكفلها القانون

بعد مناقشتها والحصول على إجابة لكل أسئلتي ، أقبل بحرية وطواعية أن أشارك في البحث الذي اقترح علي

في مراكش ،

توقيع المريض اسم وتوقيع المحقق